CLINICAL TRIAL: NCT06981338
Title: Guttmann NeuroRecovery - Viability, Safety, and Efficacy of Intrathecal Wharton's Jelly Mesenchymal Stem Cells and Transcutaneous Spinal Cord Stimulation in Chronic Spinal Cord Injury Rehabilitation: A Pilot Study
Brief Title: Guttmann NeuroRecovery - Viability, Safety, and Efficacy of Intrathecal Wharton's Jelly Mesenchymal Stem Cells and Transcutaneous Spinal Cord Stimulation in Chronic Spinal Cord Injury Rehabilitation
Acronym: GNR-SCI-01
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut Guttmann (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNR-SCI-01; 2025-521877-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-02; First posted 2025-05-20 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries (SCI); Spinal Cord Injury; Traumatic Spinal Cord Injuries; Spinal Cord Disease
Keywords: Mesenchymal Stem Cells; Spinal Cord Injuries; Cell- and Tissue-Based Therapy; Intrathecal Administration; Neuroplasticity; Spinal Cord Stimulation; Safety; Clinical Trials, Phase I; Electric Stimulation Therapy; Feasibility Study
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Intervention Model Description: This single-arm, open-label pilot study combines intrathecal Wharton's jelly mesenchymal stem cells (3 doses of 30×10⁶±30% cells at 6week-intervals) with transcutaneous spinal cord stimulation (tSCS) in chronic SCI patients (AIS A-C, 1-5 years post-injury). The model evaluates:
  * Safety (AEs, neurological/immunological monitoring)
  * Feasibility (adherence/retention rates)
  * Efficacy signals (motor/sensory/autonomic improvements via ASIA, neurophysiological tests).
  * All participants receive active treatment with 12-month core follow-up + 2-year extended safety monitoring.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic WJ-MSCs + tSCS-Assisted Neurorehabilitation (Experimental): All participants receive three intrathecal doses of allogeneic Wharton's jelly mesenchymal stem cells (30×10⁶±30% viable cells/dose) at 6-week intervals, combined with transcutaneous spinal cord stimulation (tSCS)-assisted neurorehabilitation.
  Interventions: Combination Product: Allogeneic Wharton's jelly mesenchymal stem cells (WJ-MSCs)

INTERVENTIONS:
Combination Product: Allogeneic Wharton's jelly mesenchymal stem cells (WJ-MSCs) — This experimental treatment combines intrathecal administration of allogeneic Wharton's jelly mesenchymal stem cells (WJ-MSCs) with transcutaneous spinal cord stimulation (tSCS) and neurorehabilitation. Participants will receive three doses of cryopreserved WJ-MSCs (30×10⁶±30% viable cells per dose) derived from umbilical cord tissue, delivered via lumbar puncture at 6-week intervals in a saline-albumin solution. The intervention includes concurrent tSCS, a non-invasive electrical stimulation technique, paired with standardised neurorehabilitation. As the first clinical study evaluating this specific combined therapy for chronic spinal cord injury (AIS A-C grades), safety monitoring incorporates regular cerebrospinal fluid analysis to assess potential immune responses.
  Other Names: Transcutaneous spinal cord stimulation (tSCS)

SUMMARY:
This clinical trial primarily aims to evaluate the safety and feasibility of a combined therapeutic approach for chronic spinal cord injury (SCI). The study will investigate whether the combination of intrathecal Wharton's jelly mesenchymal stem cells and transcutaneous spinal cord stimulation (tSCS) is safe and viable in individuals with chronic traumatic SCI.

The trial will enrol 10 participants aged 16-70 with traumatic SCI (cervical or thoracic levels C1-T12) classified as ASIA Impairment Scale A-C, who are 1-5 years post-injury. Participants will receive three intrathecal injections of Wharton's jelly mesenchymal stem cells, each containing 30 million viable cells (±30%), administered intrathecally at the L3-L4 level. This cellular therapy will be combined with transcutaneous spinal cord stimulation and intensive neurorehabilitation.

Participants will undergo comprehensive assessments over a 12-month follow-up period to monitor safety, feasibility, and secondarily to evaluate potential improvements in motor, sensory, and autonomic functions. Additional annual follow-up will continue for 2 years after study completion to evaluate long-term safety.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 16-70 years (parental consent required for 16-18-year-olds)
* Single traumatic spinal cord injury (AIS A-C) at C1-T12 levels
* Chronic injury (1-5 years post-injury)
* Stable medical condition with life expectancy >2 years
* Ability to attend follow-up visits and comply with all study procedures
* Written informed consent (and parental consent for minors)
* Sufficient cognitive capacity to understand the study
* For women of childbearing potential: use of effective contraception (hormonal, intrauterine device, barrier methods, sterilization, or post-menopausal status >1 year)

Exclusion Criteria:

* Severe comorbidities (e.g., cardiovascular instability, active infections)
* Individuals requiring mechanical ventilation
* Contraindications for tSCS (e.g., implanted devices)
* Pregnancy or breastfeeding
* Neurodegenerative diseases
* Significant haematological/biochemical abnormalities
* Active or recent (≤5 years) malignancy without complete remission
* Positive serology for HIV, hepatitis B virus, hepatitis C virus, or syphilis
* Communication barriers (language, aphasia)
* Concurrent participation in another clinical trial (within 30 days)
* Recent intrathecal medication or immunosuppressants (within 60 days)
* Multi-level spinal lesions or lesions >3 spinal segments on MRI
* Contraindications for lumbar puncture
* Planned spinal surgery within 24 months
* Inability to participate in rehabilitation
* Known allergies to stem cell preparation components

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) in Chronic SCI | Baseline through Month 12 post-treatment
  Safety assessment evaluating:
  1. Neurological worsening (≥1-grade decline on the American Spinal Injury Association (ASIA) Impairment Scale [AIS], grades A-E, where higher grades indicate better function).
  2. Cerebrospinal fluid (CSF) abnormalities (e.g., pleocytosis, elevated protein).
  3. Procedure-related complications (e.g., post-lumbar puncture headache, infection).
  Unit of Measure: Composite binary outcome (presence/absence of any TEAE).
Protocol Adherence Rate for Combined WJ-MSCs and tSCS Therapy | From baseline to week 18.
  Feasibility assessment measuring adherence to:
  1. Scheduled intrathecal WJ-MSC administrations (3 doses at 6-week intervals).
  2. Concomitant tSCS-assisted neurorehabilitation sessions (18 weeks). Unit of Measure: Percentage of completed interventions vs. planned (%).

SECONDARY OUTCOMES:
Change in American Spinal Injury Association (ASIA) Impairment Scale [AIS] Motor Score | Baseline to Month 12
  Change in motor function measured by the American Spinal Injury Association (ASIA) Impairment Scale [AIS] Motor Score, which evaluates voluntary muscle strength across 10 key muscle groups (0-5 points per muscle, total range 0-100). Higher scores indicate better motor function.
  Unit of Measure: Points on American Spinal Injury Association (ASIA) Impairment Scale [AIS] Motor Scale.
Change in American Spinal Injury Association (ASIA) Impairment Scale [AIS] Light Touch Sensory Score | Baseline to Month 12.
  Change in light touch sensation measured by the American Spinal Injury Association (ASIA) Impairment Scale [AIS] Light Touch Sensory Score (0-112 points, tested across 28 dermatomes). Higher scores indicate better sensory function.
  Unit of Measure: Points on American Spinal Injury Association (ASIA) Impairment Scale [AIS] Light Touch Scale.
Change in American Spinal Injury Association (ASIA) Impairment Scale [AIS] Pinprick Sensory Score | Baseline to Month 12.
  Change in pinprick sensation measured by the American Spinal Injury Association (ASIA) Impairment Scale [AIS] Pinprick Sensory Score (0-112 points, tested across 28 dermatomes). Higher scores indicate better sensory function.
  Unit of Measure: Points on American Spinal Injury Association (ASIA) Impairment Scale [AIS] Pinprick Scale.
Change in Autonomic Control | Baseline to Month 12.
  Change in autonomic function (e.g., bladder, bowel, cardiovascular regulation) assessed using the International Standards to document Autonomic Function after Spinal Cord Injury (ISAFSCI). Scores range from 0 (no function) to 2 (normal function) per domain. Higher scores indicate better autonomic control.
  Unit of Measure: Autonomic Function after Spinal Cord Injury (ISAFSCI) composite score.
Change in Motor Evoked Potential (MEP) Amplitude | Baseline to Month 12.
  Change in corticospinal tract integrity measured by Motor Evoked Potential (MEP) amplitude during transcranial magnetic stimulation. In the absence of pathological hyperexcitability, higher MEP amplitudes generally reflect better corticospinal tract integrity.
  Unit of Measure: Microvolts (µV).
Change in Motor Evoked Potential (MEP) Latency | Baseline to Month 12.
  Change in corticospinal conduction speed measured by Motor Evoked Potential (MEP) latency during transcranial magnetic stimulation. Shorter latencies generally reflect faster, more efficient corticospinal tract conduction.
  Unit of Measure: Milliseconds (ms).
Change in Somatosensory Evoked Potential (SSEP) Amplitude | Baseline to Month 12.
  Change in dorsal column-medial lemniscus pathway integrity measured by Somatosensory Evoked Potential (SSEP) amplitude during peripheral nerve stimulation. In the absence of pathological hyperexcitability, higher SSEP amplitudes generally reflect better somatosensory pathway integrity.
  Unit of Measure: Microvolts (µV).
Change in Somatosensory Evoked Potential (SSEP) Latency | Baseline to Month 12.
  Change in somatosensory pathway conduction speed measured by Somatosensory Evoked Potential (SSEP) latency during peripheral nerve stimulation. Shorter latencies generally reflect faster, more efficient conduction along the dorsal column-medial lemniscus pathway.
  Unit of Measure: Milliseconds (ms).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Guttmann: Hospital de Neurorehabilitació, Badalona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No